CLINICAL TRIAL: NCT02036814
Title: A PROGRAM OF HEALTH EDUCATION PROMOTION BY NURSING CAN IMPROVE BLOOD PRESSURE CONTROL AND QUALITY OF LIFE IN HYPERTENSIVE PATIENTS?
Brief Title: Program for Health Promotion to Improve Therapeutic Compliance in Hypertensive Patiente
Acronym: PHPTCHP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: InCor Heart Institute (Other)
Responsible Party: Principal Investigator, Grazia Maria Guerra, Grazia M. Guerra, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: CAPPesq779/05
Record Dates: First submitted 2013-10-11; First posted 2014-01-15 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2014-01

CONDITIONS: Hypertension
Keywords: Hypertension; Nursing; Therapeutic compliance; Quality of life; Health education
MeSH Terms: conditions — Hypertension; Patient Compliance; Health Education

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A who underwent to an inter-relational strategy (Experimental): Group A who underwent to a health educational orientation program (inter-relational strategy)
  Interventions: Behavioral: Program Health Education
- Group B who underwent group orientation by the nurse (Experimental)
  Interventions: Behavioral: Program Health Education

INTERVENTIONS:
Behavioral: Program Health Education

SUMMARY:
The aim was to test if interpersonal relationships group strategies provided by nursing can promote an additional benefit on blood pressure (BP) control and quality of life (QoL) in hypertensive patients. Methods: 21 treated patients were randomized into two groups: Group A 10 patients (8 women), underwent to a health educational orientation program (inter-relational strategy), with group meetings every 15 days during 4 months(8 meetings). Group B 11 patients (7 women), who underwent group orientation by the nurse every 40 days during 4 months (3 meetings). Both groups received the same content guidelines (healthy lifestyle and prevention of risk factors). The patients had 2 visits by nurses at baseline (15 days) and at the final study (120 days). BP was measured by auscultatory method and QoL questionnaire (WHOQoL-Brief)was applied. The dispensing and pill counts were done every 30 days. Ambulatory blood pressure monitoring (ABPM) was performed at baseline and after 120 days.

ELIGIBILITY:
Inclusion criteria:

* Hypertensive patients under treatment regimen;
* Pressure levels greater than or equal to 90 mmHg diastolic blood pressure (DBP), and
* Pressure level greater than or equal to 140 mmHg systolic blood pressure (SBP)
* Age limit between 25 to 75 years, for both female and male.

Exclusion Criteria:

* Diabetes patients

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
measure blood pressure arterial | 4 months
  At the first nurse interview (day 0: randomization) three consecutive measurements of BP were taken after the patient had rested for 5 min in the supine position.Ambulatory BP monitoring was recorded at 15 and 180 days of follow-up for 24 h with a noninvasive ABPM (Space Labs 90207 monitor; Space Labs, Redmond, WA) with an appropriate-sized cuff. The monitor was placed on the nondominant arm and was set to take BP readings every 10 min during the day and every 20 min at night

SECONDARY OUTCOMES:
QoL questionnaire (WHOQoL-Brief) | 4 months
  At the first nurse interview (day 0: randomization), a questionnaire was used to obtain information related to general data, habits, history of disease, other risk factors for cardiovascular disease, and prescribed medications. This questionnaire was used only to characterize the adherence behavior and the risk factors at the beginning the study, but was not used to evaluate modifications of behavior during the study.

CONTACTS AND LOCATIONS:
Overall Officials: Heno Ferreira Lopes, PhD, Study Chair — Heart Institute of Medicine School of University of São Paulo